CLINICAL TRIAL: NCT05768178
Title: DETERMINE (Determining Extended Therapeutic Indications for Existing Drugs in Rare Molecularly Defined Indications Using a National Evaluation Platform Trial): An Umbrella-Basket Platform Trial to Evaluate the Efficacy of Targeted Therapies in Rare Adult, Paediatric and Teenage/Young Adult (TYA) Cancers With Actionable Genomic Alterations, Including Common Cancers With Rare Actionable Alterations. Treatment Arm 05: Vemurafenib in Combination With Cobimetinib in Adult Patients With BRAF Positive Cancers.
Brief Title: DETERMINE Trial Treatment Arm 05: Vemurafenib in Combination With Cobimetinib in Adult Patients With BRAF Positive Cancers.
Acronym: DETERMINE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: University of Manchester (Other); University of Birmingham (Other); Royal Marsden NHS Foundation Trust (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/21/004 - Treatment Arm 5; IRAS ID: 1004057 (Other: IRAS)
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Haematological Malignancy; Melanoma; Thyroid Cancer, Papillary; Ovarian Neoplasms; Colorectal Neoplasms; Laryngeal Neoplasms; Carcinoma, Non-Small-Cell Lung; Glioma; Multiple Myeloma; Erdheim-Chester Disease; Thyroid Carcinoma, Anaplastic; Solid Tumour
Keywords: Adult; Antineoplastic Agents; Cancer; Malignancy; Malignant Neoplasms; Molecular Targeted Therapy; Mutation; Neoplasms by Histologic Type; Neoplasms by Site; Precision Medicine; Cobimetinib; Proto-Oncogene Proteins B-raf; Rare; Tumour-agnostic; Vemurafenib
MeSH Terms: conditions — Hematologic Neoplasms; Melanoma; Thyroid Cancer, Papillary; Ovarian Neoplasms; Colorectal Neoplasms; Laryngeal Neoplasms; Carcinoma, Non-Small-Cell Lung; Glioma; Multiple Myeloma; Erdheim-Chester Disease; Thyroid Carcinoma, Anaplastic; Neoplasms; Neoplasms by Histologic Type; Neoplasms by Site | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm 05 - Vemurafenib and Cobimetinib (Experimental): This vemurafenib and cobimetinib treatment arm is for BRAF V600 mutation-positive cancers occurring in adults.
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: Vemurafenib — Patients will receive vemurafenib at a dose of 960 mg orally (four tablets of 240 mg) on a twice daily schedule throughout a 28-day cycle. Patients may continue until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Zelboraf
Drug: Cobimetinib — Patients will receive cobimetinib at a dose of 60 mg (three tablets of 20 mg) to be taken orally, once daily for 21 consecutive days (days 1 to 21 in each 28-day cycle); followed by a 7-day break. Patients may continue until disease progression without clinical benefit, unacceptable AEs or withdrawal of consent.
  Other Names: Cotellic

SUMMARY:
This clinical trial is looking at a combination of drugs called vemurafenib and cobimetinib. Vemurafenib is approved as standard of care for adult patients with unresectable or metastatic melanoma. Cobimetinib is approved as standard of care in combination with vemurafenib for the treatment of adult patients with unresectable or metastatic melanoma. This means it has gone through clinical trials and been approved by the Medicines and Healthcare products Regulatory Agency (MHRA) in the UK.

Cobimetinib and vemurafenib work in patients with these types of cancers which have certain changes in the cancer cells called BRAF V600 mutation-positive.

Investigators now wish to find out if it will be useful in treating patients with other cancer types which are also BRAF V600 mutation-positive. If the results are positive, the study team will work with the NHS and the Cancer Drugs Fund to see if these drugs can be routinely accessed for patients in the future.

This trial is part of a trial programme called DETERMINE. The programme will also look at other anti-cancer drugs in the same way, through matching the drug to rare cancer types or ones with specific mutations.

DETAILED DESCRIPTION:
DETERMINE Treatment Arm 05 (vemurafenib and cobimetinib) aims to evaluate the efficacy of vemurafenib and cobimetinib in adult patients with rare* cancers with BRAF V600 mutations or in common cancers where BRAF V600 mutations are considered to be infrequent.

*Rare is defined generally as incidence less than 6 cases in 100,000 patients or common cancers with rare alterations.

This treatment arm has a target sample size of 30 evaluable patients. Sub-cohorts may be defined and further expanded to a target of 30 evaluable patients each.

The ultimate aim is to translate positive clinical findings to the NHS (Cancer Drugs Fund) to provide new treatment options for rare adult cancers.

OUTLINE:

Pre-screening: The Molecular Tumour Board makes a treatment recommendation for the patient based on molecularly-defined cohorts.

Screening: Consenting patients undergo biopsy and collection of blood samples for research purposes.

Treatment: Patients will receive vemurafenib and cobimetinib until disease progression without clinical benefit, unacceptable adverse events (AEs) or withdrawal of consent. Patients will also undergo collection of blood samples at various intervals while receiving treatment and at End of Treatment (EoT).

After completion of study treatment, patients are followed up every 3 months for 2 years.

THE DETERMINE TRIAL MASTER (SCREENING) PROTOCOL:

Please see DETERMINE Trial Master (Screening) Protocol record (NCT05722886) for information on the DETERMINE Trial Master Protocol and applicable documents.

ELIGIBILITY:
THE PATIENT MUST FULFIL THE ELIGIBILITY CRITERIA WITHIN THE DETERMINE MASTER PROTOCOL (NCT05722886) AND WITHIN THE TREATMENT ARM 05 (VEMURAFENIB AND COBIMETINIB) OUTLINED BELOW*

*When vemurafenib and cobimetinib-specific inclusion/exclusion criteria or precautions below differ from those specified in the Master Protocol, the vemurafenib and cobimetinib-specific criteria will take precedence.

Inclusion Criteria:

A. Confirmed diagnosis of a malignancy harbouring any actionable BRAF V600 mutation using an analytically validated next-generation sequencing method.

B. Adult patients ≥18 years old.

C. Patients must be able and willing to undergo a fresh tissue biopsy at baseline and blood samples for translational research. Note that for patients with haematological malignancies or neuroblastomas, blood, bone marrow aspiration and/or trephine or lymph node biopsy samples may be taken.

D. Adequate organ function as per haematological and biochemical indices within the ranges defined in the protocol. These measurements should be performed to confirm the patient's eligibility.

E. Women of childbearing potential are eligible provided that they meet the following criteria:

* Have a negative serum or urine pregnancy test before enrolment and;
* Agree to sexual abstinence OR to use any two forms of highly effective or effective methods together (at least one to be non-hormonal) such as:

  * Highly effective methods:
* combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* intrauterine device (IUD)
* intrauterine hormone-releasing system (IUS)
* bilateral tubal occlusion
* vasectomised partner

  * Effective methods:
* progestogen-only oral hormonal contraception not associated with inhibition of ovulation
* male or female condom with or without spermicide
* cap, diaphragm or sponge with spermicide

Effective from the first administration of vemurafenib or cobimetinib (whichever is first), throughout the trial and for six months after the last administration of vemurafenib or cobimetinib (whichever is later).

F. Male patients with partners who are women of childbearing potential, are eligible provided that they agree to the following, from the first administration of vemurafenib or cobimetinib (whichever is first), throughout the trial and for six months after the last administration of vemurafenib or cobimetinib (whichever is later):

* Agree to take measures not to father children by using a barrier method of contraception (condom plus spermicide) or to sexual abstinence
* Non-vasectomised male patients with partners who are women of childbearing potential must also be willing to ensure that their partner uses a highly effective method of contraception as in E, above.
* Male patients with pregnant or lactating partners must be advised to use barrier method contraception (e.g. condom) to prevent drug exposure of the foetus or neonate.

All male patients must refrain from donating sperm for the same period.

Exclusion Criteria:

A. Diagnosis of unresectable or metastatic melanoma with a BRAF V600 mutation.

B. Female patients who are pregnant, breastfeeding or planning to become pregnant during the trial or for six months following their last dose of vemurafenib or cobimetinib, whichever is later.

C. Patients with QTcF (Corrected QT interval by Fridericia) at screening of >450 ms for males and >470 ms for females measured on triplicate ECG (if 1/3 readings show >450/470 ms then patient is ineligible).

D. Patients with any history of long QT syndrome or Torsades de Pointes (or any concurrent medication with a known risk of inducing Torsades de Pointes).

E. Known hypersensitivity to vemurafenib or cobimetinib or any of the excipients.

F. Patients unable to swallow vemurafenib and cobimetinib intact, without chewing or crushing the tablets (as per the dosing schedule).

G. Patients who were administered a live, attenuated vaccine within 28 days prior to enrolment, or anticipation of need for such a vaccine during vemurafenib and cobimetinib treatment or within six months after the final dose of vemurafenib and cobimetinib.

H. Patients with clinically significant pre-existing cardiac conditions including (within the last three months prior to screening):

* Uncontrolled or symptomatic angina,
* Uncontrolled atrial or ventricular arrhythmias,
* Class III & IV New York Heart Association congestive heart failure,
* Left ventricular ejection fraction (LVEF) <50%,
* Myocardial infarction

I. Ophthalmological disorders: History of retinal detachment, severe visual impairment, central serous chorioretinopathy, neovascular retinopathy, or retinopathy of prematurity.

Patients with low grade gliomas causing visual impairment may be considered eligible and monitored with close ophthalmological monitoring.

J. History of pancreatitis.

K. History of central nervous system (CNS) or gastrointestinal (GI) haemorrhage within three months of trial entry.

L. Patients with any history of haemorrhagic stroke.

M. Prior treatment with the same class of drug unless presence of a resistance alteration known to be potentially sensitive to either vemurafenib or cobimetinib. Prior sorafenib use is permissible following a washout period of 10 days.

N. Any clinically significant concomitant disease or condition (or its treatment) that could interfere with the conduct of the trial or absorption of oral medications that would, in the opinion of the Investigator, pose an unacceptable risk to the patient in this trial.

O. Known active infections (bacterial, fungal or viral) that would interfere with the assessment of safety or efficacy of vemurafenib and cobimetinib, including human immunodeficiency virus (HIV) positivity. Patients with history of testing positive for HIV infection are eligible provided the each of the following conditions are met:

* CD4 count ≥350/μL;
* undetectable viral load;
* receiving antiretroviral therapy (ART) that does not interact with IMP (patients should be on established ART for at least four weeks); and
* no HIV/ acquired immune deficiency syndrome-associated opportunistic infection in the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  An OR is defined as the confirmed occurrence of either a Complete Response (CR) or Partial Response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 criteria (or immune related [ir]-RECIST or standard imaging criteria for specific disease e.g. Response Evaluation in Neuro Oncology criteria [RANO]). In patients with leukaemia, OR will be defined as the occurrence of CR, CRi (CR with incomplete neutrophil recovery) or CRp (CR with incomplete platelet recovery). The trial will report the proportion of patients with an OR and 95% credible interval.
Durable Clinical Benefit (DCB) | Disease assessments to be performed up to 24 weeks from the start of trial treatment.
  DCB is defined as the absence of disease progression for at least 24 weeks from the start of trial treatment according to RECIST Version 1.1 criteria (or ir-RECIST or standard imaging criteria for specific disease e.g. RANO criteria) and, where relevant (e.g. for haematological malignancies), by standard bone marrow response assessment criteria. Alternative definitions of DCB based on different time points may be pre-specified for particular sub-cohorts if 24 weeks is not clinically relevant. The trial will report the proportion of patients with a DCB and 95% credible interval.

SECONDARY OUTCOMES:
Duration of response (DR) | Disease assessment every 2 cycles (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits occur every 3 months after last dose of vemurafenib and cobimetinib for up to 2 years.
  DR is defined as the time from the date of the first confirmed CR or PR according to RECIST 1.1 or ir-RECIST (or standard imaging criteria for specific disease e.g. RANO criteria) to the date of disease progression. The trial will report the median DR and 95% credible interval.
Best percentage change in sum of target lesion / index lesion diameters (PCSD) | Disease assessment every 2 cycles (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits occur every 3 months after last dose of vemurafenib and cobimetinib for up to 2 years.
  PCSD is defined as the greatest decrease or least increase in the sum of target lesion diameters (RECIST) or index lesion diameters (irRECIST) as a percentage compared to the baseline measurement. The trial will report the mean PCSD and 95% credible interval.
Time to treatment discontinuation (TTD) | From first dose of vemurafenib and cobimetinib to discontinuation of trial treatment up to 5 years.
  TTD is defined as the time from date of starting trial treatment to date of discontinuing trial treatment, in days estimated by the median of the posterior inverse gamma probability distribution. The trial will report the median TTD and 95% credible interval.
Progression-Free Survival time (PFS) | Disease assessment every 2 cycles (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits occur every 3 months after last dose of vemurafenib and cobimetinib for up to 2 years.
  PFS is defined as the time from date of starting trial treatment to date of progression or date of death without a previous progression recorded estimated by the median of the posterior inverse gamma probability distribution.
Time to Progression (TTP) | Disease assessment every 2 cycles (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits occur every 3 months after last dose of vemurafenib and cobimetinib for up to 2 years.
  TTP is defined as the time from date of starting trial treatment to date of progression or date of death without recorded progression censored rather than events. The trial will report the median TTP and 95% credible interval.
Growth Modulation Index (GMI) | Disease assessment every 2 cycles (each cycle is 28 days) and at EoT. After 24 weeks, it can be done every 12 weeks, on discussion with Sponsor. Follow-up visits occur every 3 months after last dose of vemurafenib and cobimetinib for up to 2 years.
  GMI is defined as the ratio of TTP with the trial protocol treatment to TTP on the most recent prior line of therapy. The trial will report the mean GMI and 95% credible interval.
Overall Survival time (OS) | Time of death or up to 2 years after the EoT visit.
  OS is defined as the time from date of starting trial treatment to date of death from any cause estimated by the median of the posterior normal probability distribution.
Occurrence of at least one Suspected Unexpected Serious Adverse Reaction (SUSAR) | From the time of consent until 28 days after last dose of vemurafenib or cobimetinib (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  The trial will report the number of patients who experience at least one SUSAR to vemurafenib and cobimetinib.
Occurrence of at least one Grade 3, 4 or 5 vemurafenib and/or cobimetinib related AE | From the time of consent until 28 days after last dose of vemurafenib or cobimetinib (up to 5 years) or until patient starts another anti-cancer therapy, whichever came first. An average time frame will be presented with results entry.
  Number of patients who experience at least one vemurafenib and/or cobimetinib related Grade 3, 4 or 5 AE according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0.
EORTC-QLQ-C30 Standardised Area Under Summary Score Curve (QLQSAUC) | QoL surveys performed prior to inclusion, every cycle (each cycle is 28 days) and at EoT visit (up to 5 years).
  Multiple measures of Quality of Life (QoL) will be generated from patient completion of the European Organisation for Research and Treatment of Cancer QLQ-C30 (EORTC-QLQ-C30) questionnaire (15 measures). For each patient the Summary Score from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean QLQSAUC and 95% credible interval.
EQ-5D Standardised Area Under Index Value Curve (EQ5DSAUC) | QoL surveys performed prior to inclusion, every cycle (each cycle is 28 days) and at EoT visit (up to 5 years).
  Two measures of QoL will be generated from patient completion of the EQ-5D-5L questionnaire. For each measure, scores based on responses from the questionnaire will be generated at each time point and the area under the curve generated by these scores over time will be calculated and standardised by the time frame. The trial will report the mean EQ5DSAUC and 95% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krebs, Dr, Principal Investigator — The Christie Hospital
Locations (16):
- United Kingdom (16):
  - Belfast City Hospital, Belfast
  - University Hospital Birmingham, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - The Beatson Hospital, Glasgow
  - Leicester Royal Infirmary, Leicester
  - University College London Hospital, London
  - Guy's Hospital, London
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified patient data will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All requests for data relating to this treatment arm that are made within 5 years from last patient last visit for the vemurafenib and cobimetinib treatment arm will be considered; requests made subsequently will be considered where possible.
Access Criteria: When a request has been approved, Cancer Research UK will provide access to the de-identified individual patient-level data and appropriate supporting information. A signed Data Sharing Agreement must be in place before accessing requested information. Requests should be submitted to drugdev@cancer.org.uk.

REFERENCES:
- See also: Overview of the DETERMINE trial — http://CRUK.org/determine
- See also: ClinicalTrials.gov record for DETERMINE Trial Master Screening Protocol (NCT05722886). — https://clinicaltrials.gov/ct2/show/NCT05722886